CLINICAL TRIAL: NCT03331978
Title: A Randomized Controlled Trial of an Antiretroviral Treatment Adherence Intervention for HIV+ African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01NR017334 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS
Keywords: Adherence; Antiretroviral treatment; Black/ AfricanAmerican
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rise - Treatment Education (Experimental): Rise consists of a one-month intensive intervention (with three core 60-minute counseling sessions at weeks 1, 2, and 4) followed by two booster sessions (at weeks 12 and 20). If participants show nonadherence during booster sessions, they are offered up to four additional booster sessions (i.e., extra booster sessions if <85% of prescribed doses were taken in the past month). Thus, participants receive three core sessions in the first month, followed by 2-6 booster sessions over the next four months.
  Interventions: Behavioral: Rise - Treatment Education
- Control - No Treatment Education (No Intervention): The Usual Care control group will only receive standard of care through their HIV clinics.

INTERVENTIONS:
Behavioral: Rise - Treatment Education — Rise consists of a one-month intensive intervention (with three core 60-minute counseling sessions at weeks 1, 2, and 4) followed by two booster sessions (at weeks 12 and 20). If participants show nonadherence during booster sessions, they are offered up to four additional booster sessions (i.e., extra booster sessions if <85% of prescribed doses were taken in the past month). Thus, participants receive three core sessions in the first month, followed by 2-6 booster sessions over the next four months.
  Arms: Rise - Treatment Education

SUMMARY:
Project Rise is a randomized controlled trial (RCT) of an innovative, culturally congruent treatment education (TE) intervention for African Americans with HIV that targets cultural and social issues contributing to health disparities.

DETAILED DESCRIPTION:
Project Rise is a randomized controlled trial (RCT) of an innovative, culturally congruent treatment education (TE) intervention for African Americans with HIV that targets cultural and social issues contributing to health disparities. TE facilitates patient navigation through the medical system and provides treatment education and client-centered counseling to improve adherence and retention in care. TE targets structural issues in healthcare and patients' lives by advocating to providers to improve patient-provider relationships, recommending changes in treatment and/or providers, and referring patients to mental health and social services.

A total of 350 Black participants will be recruited through APLA Health and randomly assigned to the intervention or usual care control group (175 per group). Adherence will be electronically monitored daily (and downloaded bi-monthly) from baseline to 13-months post-baseline. Viral load will be assessed through venipuncture at baseline and 6- and 13-months post-baseline. It is hypothesized that the intervention group will show better adherence and have a greater likelihood of suppressed viral load than the control group over time.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* 18 years of age or older
* Self-identified as African American/Black
* Been prescribed antiretroviral therapy (ART) in the past 12 months
* Self-reported adherence problems (i.e. missed at least 1 ART dose in the past month) and/or detectable viral load
* Willing to use Medication Events Monitoring System (MEMS) for electronic adherence monitoring.

Exclusion Criteria:

* HIV-negative
* 17 years of age or younger
* Not self-identified as African American/Black, not on antiretroviral therapy (ART) or not prescribed ART therapy in the last than 12 months
* No self-reported adherence problems and/or no detectable viral load
* Not willing to use Medication Events Monitoring System (MEMS) for electronic adherence monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AIDS Project Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simoni JM, Huh D, Wilson IB, Shen J, Goggin K, Reynolds NR, Remien RH, Rosen MI, Bangsberg DR, Liu H. Racial/Ethnic disparities in ART adherence in the United States: findings from the MACH14 study. J Acquir Immune Defic Syndr. 2012 Aug 15;60(5):466-72. doi: 10.1097/QAI.0b013e31825db0bd. PMID 22595873
- [Background] Giordano TP, Bartsch G, Zhang Y, Tedaldi E, Absalon J, Mannheimer S, Thomas A, MacArthur RD. Disparities in outcomes for African American and Latino subjects in the Flexible Initial Retrovirus Suppressive Therapies (FIRST) trial. AIDS Patient Care STDS. 2010 May;24(5):287-95. doi: 10.1089/apc.2009.0332. PMID 20438378
- [Background] Bogart LM, Bird ST, Walt LC, Delahanty DL, Figler JL. Association of stereotypes about physicians to health care satisfaction, help-seeking behavior, and adherence to treatment. Soc Sci Med. 2004 Mar;58(6):1049-58. doi: 10.1016/s0277-9536(03)00277-6. PMID 14723901
- [Background] Bogart LM, Wagner G, Galvan FH, Banks D. Conspiracy beliefs about HIV are related to antiretroviral treatment nonadherence among african american men with HIV. J Acquir Immune Defic Syndr. 2010 Apr;53(5):648-55. doi: 10.1097/QAI.0b013e3181c57dbc. PMID 19952767
- [Background] Bogart LM, Wagner GJ, Green HD Jr, Mutchler MG, Klein DJ, McDavitt B, Lawrence SJ, Hilliard CL. Medical mistrust among social network members may contribute to antiretroviral treatment nonadherence in African Americans living with HIV. Soc Sci Med. 2016 Sep;164:133-140. doi: 10.1016/j.socscimed.2016.03.028. Epub 2016 Mar 19. PMID 27046475
- [Background] Earnshaw VA, Bogart LM, Dovidio JF, Williams DR. Stigma and racial/ethnic HIV disparities: moving toward resilience. Am Psychol. 2013 May-Jun;68(4):225-36. doi: 10.1037/a0032705. PMID 23688090
- [Background] Bogart LM, Wagner GJ, Green HD Jr, Mutchler MG, Klein DJ, McDavitt B. Social Network Characteristics Moderate the Association Between Stigmatizing Attributions About HIV and Non-adherence Among Black Americans Living with HIV: a Longitudinal Assessment. Ann Behav Med. 2015 Dec;49(6):865-72. doi: 10.1007/s12160-015-9724-1. PMID 26296702
- [Background] Dale SK, Bogart LM, Wagner GJ, Galvan FH, Klein DJ. Medical mistrust is related to lower longitudinal medication adherence among African-American males with HIV. J Health Psychol. 2016 Jul;21(7):1311-21. doi: 10.1177/1359105314551950. Epub 2014 Oct 7. PMID 25293970
- [Background] Wagner GJ, Bogart LM, Galvan FH, Banks D, Klein DJ. Discrimination as a key mediator of the relationship between posttraumatic stress and HIV treatment adherence among African American men. J Behav Med. 2012 Feb;35(1):8-18. doi: 10.1007/s10865-011-9320-1. Epub 2011 Feb 12. PMID 21318411
- [Background] Bogart LM, Landrine H, Galvan FH, Wagner GJ, Klein DJ. Perceived discrimination and physical health among HIV-positive Black and Latino men who have sex with men. AIDS Behav. 2013 May;17(4):1431-41. doi: 10.1007/s10461-012-0397-5. PMID 23297084
- [Background] Fields EL, Bogart LM, Smith KC, Malebranche DJ, Ellen J, Schuster MA. HIV risk and perceptions of masculinity among young black men who have sex with men. J Adolesc Health. 2012 Mar;50(3):296-303. doi: 10.1016/j.jadohealth.2011.07.007. Epub 2011 Oct 2. PMID 22325136
- [Background] Fields EL, Bogart LM, Galvan FH, Wagner GJ, Klein DJ, Schuster MA. Association of discrimination-related trauma with sexual risk among HIV-positive African American men who have sex with men. Am J Public Health. 2013 May;103(5):875-80. doi: 10.2105/AJPH.2012.300951. Epub 2013 Mar 14. PMID 23488499
- [Background] Fields EL, Bogart LM, Smith KC, Malebranche DJ, Ellen J, Schuster MA. "I Always Felt I Had to Prove My Manhood": Homosexuality, Masculinity, Gender Role Strain, and HIV Risk Among Young Black Men Who Have Sex With Men. Am J Public Health. 2015 Jan;105(1):122-131. doi: 10.2105/AJPH.2013.301866. PMID 24832150
- [Background] Bogart LM, Galvan FH, Wagner GJ, Klein DJ. Longitudinal association of HIV conspiracy beliefs with sexual risk among black males living with HIV. AIDS Behav. 2011 Aug;15(6):1180-6. doi: 10.1007/s10461-010-9796-7. PMID 20734227
- [Background] McGuire TG, Miranda J. New evidence regarding racial and ethnic disparities in mental health: policy implications. Health Aff (Millwood). 2008 Mar-Apr;27(2):393-403. doi: 10.1377/hlthaff.27.2.393. PMID 18332495
- [Background] Rumptz MH, Tobias C, Rajabiun S, Bradford J, Cabral H, Young R, Cunningham WE. Factors associated with engaging socially marginalized HIV-positive persons in primary care. AIDS Patient Care STDS. 2007;21 Suppl 1:S30-9. doi: 10.1089/apc.2007.9989. PMID 17563288
- [Background] Cunningham WE, Andersen RM, Katz MH, Stein MD, Turner BJ, Crystal S, Zierler S, Kuromiya K, Morton SC, St Clair P, Bozzette SA, Shapiro MF. The impact of competing subsistence needs and barriers on access to medical care for persons with human immunodeficiency virus receiving care in the United States. Med Care. 1999 Dec;37(12):1270-81. doi: 10.1097/00005650-199912000-00010. PMID 10599608
- [Background] Mathes T, Pieper D, Antoine SL, Eikermann M. Adherence-enhancing interventions for highly active antiretroviral therapy in HIV-infected patients - a systematic review. HIV Med. 2013 Nov;14(10):583-95. doi: 10.1111/hiv.12051. Epub 2013 Jun 17. PMID 23773654
- [Background] Simoni JM, Amico KR, Smith L, Nelson K. Antiretroviral adherence interventions: translating research findings to the real world clinic. Curr HIV/AIDS Rep. 2010 Feb;7(1):44-51. doi: 10.1007/s11904-009-0037-5. PMID 20425057
- [Background] Amico KR, Harman JJ, Johnson BT. Efficacy of antiretroviral therapy adherence interventions: a research synthesis of trials, 1996 to 2004. J Acquir Immune Defic Syndr. 2006 Mar;41(3):285-97. doi: 10.1097/01.qai.0000197870.99196.ea. PMID 16540929
- [Background] Wagner GJ, Bogart LM, Mutchler MG, McDavitt B, Mutepfa KD, Risley B. Increasing Antiretroviral Adherence for HIV-Positive African Americans (Project Rise): A Treatment Education Intervention Protocol. JMIR Res Protoc. 2016 Mar 29;5(1):e45. doi: 10.2196/resprot.5245. PMID 27025399
- [Background] Bogart LM, Wagner GJ, Mutchler MG, Risley B, McDavitt BW, McKay T, Klein DJ. Community HIV treatment advocacy programs may support treatment adherence. AIDS Educ Prev. 2012 Feb;24(1):1-14. doi: 10.1521/aeap.2012.24.1.1. PMID 22339141
- [Background] Mutchler MG, Wagner G, Cowgill BO, McKay T, Risley B, Bogart LM. Improving HIV/AIDS care through treatment advocacy: going beyond client education to empowerment by facilitating client-provider relationships. AIDS Care. 2011 Jan;23(1):79-90. doi: 10.1080/09540121.2010.496847. PMID 21218280
- [Background] Charania MR, Marshall KJ, Lyles CM, Crepaz N, Kay LS, Koenig LJ, Weidle PJ, Purcell DW; HIV/AIDS Prevention Research Synthesis (PRS) Team. Identification of evidence-based interventions for promoting HIV medication adherence: findings from a systematic review of U.S.-based studies, 1996-2011. AIDS Behav. 2014 Apr;18(4):646-60. doi: 10.1007/s10461-013-0594-x. PMID 24043269
- [Background] Langebeek N, Nieuwkerk P. Electronic medication monitoring-informed counseling to improve adherence to combination anti-retroviral therapy and virologic treatment outcomes: a meta-analysis. Front Public Health. 2015 May 19;3:139. doi: 10.3389/fpubh.2015.00139. eCollection 2015. PMID 26042212
- [Background] Cunningham W. HIV racial disparities: time to close the gaps. Arch Intern Med. 2012 Nov 12;172(20):1599-600. doi: 10.1001/2013.jamainternmed.613. No abstract available. PMID 23044931
- [Background] Brandon DT, Isaac LA, LaVeist TA. The legacy of Tuskegee and trust in medical care: is Tuskegee responsible for race differences in mistrust of medical care? J Natl Med Assoc. 2005 Jul;97(7):951-6. PMID 16080664
- [Background] Armstrong K, McMurphy S, Dean LT, Micco E, Putt M, Halbert CH, Schwartz JS, Sankar P, Pyeritz RE, Bernhardt B, Shea JA. Differences in the patterns of health care system distrust between blacks and whites. J Gen Intern Med. 2008 Jun;23(6):827-33. doi: 10.1007/s11606-008-0561-9. Epub 2008 Feb 26. PMID 18299939
- [Background] Armstrong K, Ravenell KL, McMurphy S, Putt M. Racial/ethnic differences in physician distrust in the United States. Am J Public Health. 2007 Jul;97(7):1283-9. doi: 10.2105/AJPH.2005.080762. Epub 2007 May 30. PMID 17538069
- [Background] Chen FM, Fryer GE Jr, Phillips RL Jr, Wilson E, Pathman DE. Patients' beliefs about racism, preferences for physician race, and satisfaction with care. Ann Fam Med. 2005 Mar-Apr;3(2):138-43. doi: 10.1370/afm.282. PMID 15798040
- [Background] Hausmann LR, Jeong K, Bost JE, Ibrahim SA. Perceived discrimination in health care and health status in a racially diverse sample. Med Care. 2008 Sep;46(9):905-14. doi: 10.1097/MLR.0b013e3181792562. PMID 18725844
- [Background] LaVeist TA, Nickerson KJ, Bowie JV. Attitudes about racism, medical mistrust, and satisfaction with care among African American and white cardiac patients. Med Care Res Rev. 2000;57 Suppl 1:146-61. doi: 10.1177/1077558700057001S07. PMID 11092161
- [Background] Lillie-Blanton M, Brodie M, Rowland D, Altman D, McIntosh M. Race, ethnicity, and the health care system: public perceptions and experiences. Med Care Res Rev. 2000;57 Suppl 1:218-35. doi: 10.1177/1077558700057001S10. PMID 11092164
- [Background] Schrimshaw EW, Siegel K, Lekas HM. Changes in attitudes toward antiviral medication: a comparison of women living with HIV/AIDS in the pre-HAART and HAART Eras. AIDS Behav. 2005 Sep;9(3):267-79. doi: 10.1007/s10461-005-9001-6. PMID 16088368
- [Background] Siegel K, Karus D, Schrimshaw EW. Racial differences in attitudes toward protease inhibitors among older HIV-infected men. AIDS Care. 2000 Aug;12(4):423-34. doi: 10.1080/09540120050123828. PMID 11091775
- [Background] O'Leary A, Fisher HH, Purcell DW, Spikes PS, Gomez CA. Correlates of risk patterns and race/ethnicity among HIV-positive men who have sex with men. AIDS Behav. 2007 Sep;11(5):706-15. doi: 10.1007/s10461-006-9205-4. PMID 17295071
- [Background] Foster PP, Gaskins SW. Older African Americans' management of HIV/AIDS stigma. AIDS Care. 2009 Oct;21(10):1306-12. doi: 10.1080/09540120902803141. PMID 20024707
- [Background] Graham LF, Braithwaite K, Spikes P, Stephens CF, Edu UF. Exploring the mental health of black men who have sex with men. Community Ment Health J. 2009 Aug;45(4):272-84. doi: 10.1007/s10597-009-9186-7. Epub 2009 Mar 17. PMID 19291399
- [Background] Peterson JL, Jones KT. HIV prevention for black men who have sex with men in the United States. Am J Public Health. 2009 Jun;99(6):976-80. doi: 10.2105/AJPH.2008.143214. Epub 2009 Apr 16. PMID 19372510
- [Background] Bogart LM, Wagner GJ, Galvan FH, Klein DJ. Longitudinal relationships between antiretroviral treatment adherence and discrimination due to HIV-serostatus, race, and sexual orientation among African-American men with HIV. Ann Behav Med. 2010 Oct;40(2):184-90. doi: 10.1007/s12160-010-9200-x. PMID 20552416
- [Background] Sayles JN, Wong MD, Cunningham WE. The inability to take medications openly at home: does it help explain gender disparities in HAART use? J Womens Health (Larchmt). 2006 Mar;15(2):173-81. doi: 10.1089/jwh.2006.15.173. PMID 16536681
- [Background] Rintamaki LS, Davis TC, Skripkauskas S, Bennett CL, Wolf MS. Social stigma concerns and HIV medication adherence. AIDS Patient Care STDS. 2006 May;20(5):359-68. doi: 10.1089/apc.2006.20.359. PMID 16706710
- [Background] Vanable PA, Carey MP, Blair DC, Littlewood RA. Impact of HIV-related stigma on health behaviors and psychological adjustment among HIV-positive men and women. AIDS Behav. 2006 Sep;10(5):473-82. doi: 10.1007/s10461-006-9099-1. PMID 16604295
- [Background] Sayles JN, Wong MD, Kinsler JJ, Martins D, Cunningham WE. The association of stigma with self-reported access to medical care and antiretroviral therapy adherence in persons living with HIV/AIDS. J Gen Intern Med. 2009 Oct;24(10):1101-8. doi: 10.1007/s11606-009-1068-8. Epub 2009 Aug 4. PMID 19653047
- [Background] Smith R, Rossetto K, Peterson BL. A meta-analysis of disclosure of one's HIV-positive status, stigma and social support. AIDS Care. 2008 Nov;20(10):1266-75. doi: 10.1080/09540120801926977. PMID 18608080
- [Background] Katz IT, Ryu AE, Onuegbu AG, Psaros C, Weiser SD, Bangsberg DR, Tsai AC. Impact of HIV-related stigma on treatment adherence: systematic review and meta-synthesis. J Int AIDS Soc. 2013 Nov 13;16(3 Suppl 2):18640. doi: 10.7448/IAS.16.3.18640. PMID 24242258
- [Background] Clark R, Anderson NB, Clark VR, Williams DR. Racism as a stressor for African Americans. A biopsychosocial model. Am Psychol. 1999 Oct;54(10):805-16. doi: 10.1037//0003-066x.54.10.805. PMID 10540593
- [Background] Smith SM, Stinson FS, Dawson DA, Goldstein R, Huang B, Grant BF. Race/ethnic differences in the prevalence and co-occurrence of substance use disorders and independent mood and anxiety disorders: Results from the National Epidemiologic Survey on Alcohol and Related Conditions. Psychol Med. 2006 Jul;36(7):987-98. doi: 10.1017/S0033291706007690. Epub 2006 May 2. PMID 16650344
- [Background] Williams DR, Gonzalez HM, Neighbors H, Nesse R, Abelson JM, Sweetman J, Jackson JS. Prevalence and distribution of major depressive disorder in African Americans, Caribbean blacks, and non-Hispanic whites: results from the National Survey of American Life. Arch Gen Psychiatry. 2007 Mar;64(3):305-15. doi: 10.1001/archpsyc.64.3.305. PMID 17339519
- [Background] Knowlton AR, Hoover DR, Chung SE, Celentano DD, Vlahov D, Latkin CA. Access to medical care and service utilization among injection drug users with HIV/AIDS. Drug Alcohol Depend. 2001 Sep 1;64(1):55-62. doi: 10.1016/s0376-8716(00)00228-3. PMID 11470341
- [Background] Naar-King S, Bradford J, Coleman S, Green-Jones M, Cabral H, Tobias C. Retention in care of persons newly diagnosed with HIV: outcomes of the Outreach Initiative. AIDS Patient Care STDS. 2007;21 Suppl 1:S40-8. doi: 10.1089/apc.2007.9988. PMID 17563289
- [Background] Shapiro MF, Morton SC, McCaffrey DF, Senterfitt JW, Fleishman JA, Perlman JF, Athey LA, Keesey JW, Goldman DP, Berry SH, Bozzette SA. Variations in the care of HIV-infected adults in the United States: results from the HIV Cost and Services Utilization Study. JAMA. 1999 Jun 23-30;281(24):2305-15. doi: 10.1001/jama.281.24.2305. PMID 10386555
- [Background] Tobias C, Cunningham WE, Cunningham CO, Pounds MB. Making the connection: the importance of engagement and retention in HIV medical care. AIDS Patient Care STDS. 2007;21 Suppl 1:S3-8. doi: 10.1089/apc.2007.9992. PMID 17563287
- [Background] Fogarty L, Roter D, Larson S, Burke J, Gillespie J, Levy R. Patient adherence to HIV medication regimens: a review of published and abstract reports. Patient Educ Couns. 2002 Feb;46(2):93-108. doi: 10.1016/s0738-3991(01)00219-1. PMID 11867239
- [Background] Boarts JM, Sledjeski EM, Bogart LM, Delahanty DL. The differential impact of PTSD and depression on HIV disease markers and adherence to HAART in people living with HIV. AIDS Behav. 2006 May;10(3):253-61. doi: 10.1007/s10461-006-9069-7. PMID 16482405
- [Background] Kidder DP, Wolitski RJ, Campsmith ML, Nakamura GV. Health status, health care use, medication use, and medication adherence among homeless and housed people living with HIV/AIDS. Am J Public Health. 2007 Dec;97(12):2238-45. doi: 10.2105/AJPH.2006.090209. Epub 2007 Oct 30. PMID 17971562
- [Background] Leaver CA, Bargh G, Dunn JR, Hwang SW. The effects of housing status on health-related outcomes in people living with HIV: a systematic review of the literature. AIDS Behav. 2007 Nov;11(6 Suppl):85-100. doi: 10.1007/s10461-007-9246-3. Epub 2007 Aug 8. PMID 17682940
- [Background] Uthman OA, Magidson JF, Safren SA, Nachega JB. Depression and adherence to antiretroviral therapy in low-, middle- and high-income countries: a systematic review and meta-analysis. Curr HIV/AIDS Rep. 2014 Sep;11(3):291-307. doi: 10.1007/s11904-014-0220-1. PMID 25038748
- [Background] Gonzalez JS, Batchelder AW, Psaros C, Safren SA. Depression and HIV/AIDS treatment nonadherence: a review and meta-analysis. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):181-7. doi: 10.1097/QAI.0b013e31822d490a. PMID 21857529
- [Background] Rosen MI, Black AC, Arnsten JH, Goggin K, Remien RH, Simoni JM, Golin CE, Bangsberg DR, Liu H. Association between use of specific drugs and antiretroviral adherence: findings from MACH 14. AIDS Behav. 2013 Jan;17(1):142-7. doi: 10.1007/s10461-011-0124-7. PMID 22246513
- [Background] Young S, Wheeler AC, McCoy SI, Weiser SD. A review of the role of food insecurity in adherence to care and treatment among adult and pediatric populations living with HIV and AIDS. AIDS Behav. 2014 Oct;18 Suppl 5(0 5):S505-15. doi: 10.1007/s10461-013-0547-4. PMID 23842717
- [Background] Katz MH, Cunningham WE, Fleishman JA, Andersen RM, Kellogg T, Bozzette SA, Shapiro MF. Effect of case management on unmet needs and utilization of medical care and medications among HIV-infected persons. Ann Intern Med. 2001 Oct 16;135(8 Pt 1):557-65. doi: 10.7326/0003-4819-135-8_part_1-200110160-00006. PMID 11601927
- [Background] Ashman JJ, Conviser R, Pounds MB. Associations between HIV-positive individuals' receipt of ancillary services and medical care receipt and retention. AIDS Care. 2002 Aug;14 Suppl 1:S109-18. doi: 10.1080/09540120220149993a. PMID 12204145
- [Background] Chan D, Absher D, Sabatier S. Recipients in need of ancillary services and their receipt of HIV medical care in California. AIDS Care. 2002 Aug;14 Suppl 1:S73-83. doi: 10.1080/0954012021000009665. PMID 12204143
- [Background] Gardner LI, Metsch LR, Anderson-Mahoney P, Loughlin AM, del Rio C, Strathdee S, Sansom SL, Siegal HA, Greenberg AE, Holmberg SD; Antiretroviral Treatment and Access Study Study Group. Efficacy of a brief case management intervention to link recently diagnosed HIV-infected persons to care. AIDS. 2005 Mar 4;19(4):423-31. doi: 10.1097/01.aids.0000161772.51900.eb. PMID 15750396
- [Background] Magnus M, Schmidt N, Kirkhart K, Schieffelin C, Fuchs N, Brown B, Kissinger PJ. Association between ancillary services and clinical and behavioral outcomes among HIV-infected women. AIDS Patient Care STDS. 2001 Mar;15(3):137-45. doi: 10.1089/108729101750123607. PMID 11313026
- [Background] Messeri PA, Abramson DM, Aidala AA, Lee F, Lee G. The impact of ancillary HIV services on engagement in medical care in New York City. AIDS Care. 2002 Aug;14 Suppl 1:S15-29. doi: 10.1080/09540120220149948. PMID 12204139
- [Background] Sherer R, Stieglitz K, Narra J, Jasek J, Green L, Moore B, Shott S, Cohen M. HIV multidisciplinary teams work: support services improve access to and retention in HIV primary care. AIDS Care. 2002 Aug;14 Suppl 1:S31-44. doi: 10.1080/09540120220149975. PMID 12204140
- [Background] Conviser R, Pounds MB. The role of ancillary services in client-centred systems of care. AIDS Care. 2002 Aug;14 Suppl 1:S119-31. doi: 10.1080/09540120220150018. PMID 12204146
- [Background] Lo W, MacGovern T, Bradford J. Association of ancillary services with primary care utilization and retention for patients with HIV/AIDS. AIDS Care. 2002 Aug;14 Suppl 1:S45-57. doi: 10.1080/0954012022014992049984. PMID 12204141
- [Background] HIV/AIDS Treatment Adherence, Health Outcomes and Cost Study Group. The HIV/AIDS Treatment Adherence, Health Outcomes and Cost Study: conceptual foundations and overview. AIDS Care. 2004;16 Suppl 1:S6-21. doi: 10.1080/09540120412331315312. PMID 15739266
- [Background] Simoni JM, Pearson CR, Pantalone DW, Marks G, Crepaz N. Efficacy of interventions in improving highly active antiretroviral therapy adherence and HIV-1 RNA viral load. A meta-analytic review of randomized controlled trials. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1(0 1):S23-35. doi: 10.1097/01.qai.0000248342.05438.52. PMID 17133201
- [Background] Goldie SJ, Paltiel AD, Weinstein MC, Losina E, Seage GR 3rd, Kimmel AD, Walensky RP, Sax PE, Freedberg KA. Projecting the cost-effectiveness of adherence interventions in persons with human immunodeficiency virus infection. Am J Med. 2003 Dec 1;115(8):632-41. doi: 10.1016/j.amjmed.2003.07.007. PMID 14656616
- [Background] Freedberg KA, Hirschhorn LR, Schackman BR, Wolf LL, Martin LA, Weinstein MC, Goldin S, Paltiel AD, Katz C, Goldie SJ, Losina E. Cost-effectiveness of an intervention to improve adherence to antiretroviral therapy in HIV-infected patients. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1:S113-8. doi: 10.1097/01.qai.0000248334.52072.25. PMID 17133193
- [Background] Schackman BR, Finkelstein R, Neukermans CP, Lewis L, Eldred L; CENTER FOR ADHERENCE SUPPORT AND EVALUATION (CASE) TEAM. The cost of HIV medication adherence support interventions: results of a cross-site evaluation. AIDS Care. 2005 Nov;17(8):927-37. doi: 10.1080/09540120500100635. PMID 16265786
- [Background] Oberje EJ, de Kinderen RJ, Evers SM, van Woerkum CM, de Bruin M. Cost effectiveness of medication adherence-enhancing interventions: a systematic review of trial-based economic evaluations. Pharmacoeconomics. 2013 Dec;31(12):1155-68. doi: 10.1007/s40273-013-0108-8. PMID 24222477
- [Background] Kaufman MR, Cornish F, Zimmerman RS, Johnson BT. Health behavior change models for HIV prevention and AIDS care: practical recommendations for a multi-level approach. J Acquir Immune Defic Syndr. 2014 Aug 15;66 Suppl 3(Suppl 3):S250-8. doi: 10.1097/QAI.0000000000000236. PMID 25007194
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Fisher JD, Amico KR, Fisher WA, Harman JJ. The information-motivation-behavioral skills model of antiretroviral adherence and its applications. Curr HIV/AIDS Rep. 2008 Nov;5(4):193-203. doi: 10.1007/s11904-008-0028-y. PMID 18838059
- [Background] Amico KR, Barta W, Konkle-Parker DJ, Fisher JD, Cornman DH, Shuper PA, Fisher WA. The information-motivation-behavioral skills model of ART adherence in a Deep South HIV+ clinic sample. AIDS Behav. 2009 Feb;13(1):66-75. doi: 10.1007/s10461-007-9311-y. Epub 2007 Sep 18. PMID 17876697
- [Background] Amico KR, Toro-Alfonso J, Fisher JD. An empirical test of the information, motivation and behavioral skills model of antiretroviral therapy adherence. AIDS Care. 2005 Aug;17(6):661-73. doi: 10.1080/09540120500038058. PMID 16036253
- [Background] Starace F, Massa A, Amico KR, Fisher JD. Adherence to antiretroviral therapy: an empirical test of the information-motivation-behavioral skills model. Health Psychol. 2006 Mar;25(2):153-62. doi: 10.1037/0278-6133.25.2.153. PMID 16569106
- [Background] Kalichman SC, Rompa D, DiFonzo K, Simpson D, Austin J, Luke W, Kyomugisha F, Buckles J. HIV treatment adherence in women living with HIV/AIDS: research based on the Information-Motivation-Behavioral Skills model of health behavior. J Assoc Nurses AIDS Care. 2001 Jul-Aug;12(4):58-67. doi: 10.1016/S1055-3290(06)60217-3. PMID 11486721
- [Background] Williams JK, Wyatt GE, Wingood G. The four Cs of HIV prevention with African Americans: crisis, condoms, culture, and community. Curr HIV/AIDS Rep. 2010 Nov;7(4):185-93. doi: 10.1007/s11904-010-0058-0. PMID 20730512
- [Background] Wyatt GE. Enhancing cultural and contextual intervention strategies to reduce HIV/AIDS among African Americans. Am J Public Health. 2009 Nov;99(11):1941-5. doi: 10.2105/AJPH.2008.152181. Epub 2009 Sep 17. PMID 19762666
- [Background] Chaiyachati KH, Ogbuoji O, Price M, Suthar AB, Negussie EK, Barnighausen T. Interventions to improve adherence to antiretroviral therapy: a rapid systematic review. AIDS. 2014 Mar;28 Suppl 2:S187-204. doi: 10.1097/QAD.0000000000000252. PMID 24849479
- [Background] Bogart LM, Wagner GJ, Galvan FH, Landrine H, Klein DJ, Sticklor LA. Perceived discrimination and mental health symptoms among Black men with HIV. Cultur Divers Ethnic Minor Psychol. 2011 Jul;17(3):295-302. doi: 10.1037/a0024056. PMID 21787061
- [Background] McDavitt B, Mutchler MG. "Dude, You're Such a Slut!" Barriers and Facilitators of Sexual Communication Among Young Gay Men and Their Best Friends. J Adolesc Res. 2014 Jul;29(4):464-498. doi: 10.1177/0743558414528974. PMID 25419044
- [Background] Mutchler MG, McDavitt B, Ghani MA, Nogg K, Winder TJ, Soto JK. Getting PrEPared for HIV Prevention Navigation: Young Black Gay Men Talk About HIV Prevention in the Biomedical Era. AIDS Patient Care STDS. 2015 Sep;29(9):490-502. doi: 10.1089/apc.2015.0002. Epub 2015 Jun 29. PMID 26121564
- [Background] McDavitt B, Bogart LM, Mutchler MG, Wagner GJ, Green HD Jr, Lawrence SJ, Mutepfa KD, Nogg KA. Dissemination as Dialogue: Building Trust and Sharing Research Findings Through Community Engagement. Prev Chronic Dis. 2016 Mar 17;13:E38. doi: 10.5888/pcd13.150473. PMID 26986541
- [Background] Bing EG, Bingham T, Millett GA. Research needed to more effectively combat HIV among African-American men who have sex with men. J Natl Med Assoc. 2008 Jan;100(1):52-6. doi: 10.1016/s0027-9684(15)31174-3. PMID 18277808
- [Background] Wagner GJ, Kanouse DE, Golinelli D, Miller LG, Daar ES, Witt MD, Diamond C, Tilles JG, Kemper CA, Larsen R, Goicoechea M, Haubrich RH. Cognitive-behavioral intervention to enhance adherence to antiretroviral therapy: a randomized controlled trial (CCTG 578). AIDS. 2006 Jun 12;20(9):1295-302. doi: 10.1097/01.aids.0000232238.28415.d2. PMID 16816559
- [Background] Wagner GJ, Lovely P, Schneider S. Pilot controlled trial of the adherence readiness program: an intervention to assess and sustain HIV antiretroviral adherence readiness. AIDS Behav. 2013 Nov;17(9):3059-65. doi: 10.1007/s10461-013-0550-9. PMID 23904145
- [Background] Wagner GJ, Ghosh-Dastidar B. Electronic monitoring: adherence assessment or intervention? HIV Clin Trials. 2002 Jan-Feb;3(1):45-51. doi: 10.1310/XGXU-FUDK-A9QT-MPTF. PMID 11819185
- [Background] Wagner GJ, Kanouse DE. Assessing usual care in clinical trials of adherence interventions for highly active antiretroviral therapy. J Acquir Immune Defic Syndr. 2003 Jun 1;33(2):276-7. doi: 10.1097/00126334-200306010-00026. No abstract available. PMID 12794566
- [Background] Cunningham WE, Hays RD, Williams KW, Beck KC, Dixon WJ, Shapiro MF. Access to medical care and health-related quality of life for low-income persons with symptomatic human immunodeficiency virus. Med Care. 1995 Jul;33(7):739-54. doi: 10.1097/00005650-199507000-00009. PMID 7596212
- [Background] Andersen R, Bozzette S, Shapiro M, St Clair P, Morton S, Crystal S, Goldman D, Wenger N, Gifford A, Leibowitz A, Asch S, Berry S, Nakazono T, Heslin K, Cunningham W. Access of vulnerable groups to antiretroviral therapy among persons in care for HIV disease in the United States. HCSUS Consortium. HIV Cost and Services Utilization Study. Health Serv Res. 2000 Jun;35(2):389-416. PMID 10857469
- [Background] Cunningham WE, Markson LE, Andersen RM, Crystal SH, Fleishman JA, Golin C, Gifford A, Liu HH, Nakazono TT, Morton S, Bozzette SA, Shapiro MF, Wenger NS. Prevalence and predictors of highly active antiretroviral therapy use in patients with HIV infection in the united states. HCSUS Consortium. HIV Cost and Services Utilization. J Acquir Immune Defic Syndr. 2000 Oct 1;25(2):115-23. doi: 10.1097/00042560-200010010-00005. PMID 11103041
- [Background] Cabral HJ, Tobias C, Rajabiun S, Sohler N, Cunningham C, Wong M, Cunningham W. Outreach program contacts: do they increase the likelihood of engagement and retention in HIV primary care for hard-to-reach patients? AIDS Patient Care STDS. 2007;21 Suppl 1:S59-67. doi: 10.1089/apc.2007.9986. PMID 17563291
- [Background] Bradford JB, Coleman S, Cunningham W. HIV System Navigation: an emerging model to improve HIV care access. AIDS Patient Care STDS. 2007;21 Suppl 1:S49-58. doi: 10.1089/apc.2007.9987. PMID 17563290
- [Background] Cunningham WE, Sohler NL, Tobias C, Drainoni ML, Bradford J, Davis C, Cabral HJ, Cunningham CO, Eldred L, Wong MD. Health services utilization for people with HIV infection: comparison of a population targeted for outreach with the U.S. population in care. Med Care. 2006 Nov;44(11):1038-47. doi: 10.1097/01.mlr.0000242942.17968.69. PMID 17063136
- [Background] Zingmond DS, Ettner SL, Cunningham WE. The impact of managed care on access to highly active antiretroviral therapy and on outcomes among Medicaid beneficiaries with AIDS. Med Care Res Rev. 2007 Feb;64(1):66-82. doi: 10.1177/1077558706296243. PMID 17213458
- [Background] Goggin K, Gerkovich MM, Williams KB, Banderas JW, Catley D, Berkley-Patton J, Wagner GJ, Stanford J, Neville S, Kumar VK, Bamberger DM, Clough LA. A randomized controlled trial examining the efficacy of motivational counseling with observed therapy for antiretroviral therapy adherence. AIDS Behav. 2013 Jul;17(6):1992-2001. doi: 10.1007/s10461-013-0467-3. PMID 23568228
- [Background] Catley D, Goggin K, Harris KJ, Richter KP, Williams K, Patten C, Resnicow K, Ellerbeck EF, Bradley-Ewing A, Lee HS, Moreno JL, Grobe JE. A Randomized Trial of Motivational Interviewing: Cessation Induction Among Smokers With Low Desire to Quit. Am J Prev Med. 2016 May;50(5):573-583. doi: 10.1016/j.amepre.2015.10.013. Epub 2015 Dec 23. PMID 26711164
- [Background] Linnemayr S, Stecher C. Behavioral Economics Matters for HIV Research: The Impact of Behavioral Biases on Adherence to Antiretrovirals (ARVs). AIDS Behav. 2015 Nov;19(11):2069-75. doi: 10.1007/s10461-015-1076-0. PMID 25987190
- [Background] Linnemayr S, Rice T. Insights From Behavioral Economics to Design More Effective Incentives for Improving Chronic Health Behaviors, With an Application to Adherence to Antiretrovirals. J Acquir Immune Defic Syndr. 2016 Jun 1;72(2):e50-2. doi: 10.1097/QAI.0000000000000972. No abstract available. PMID 26918543
- [Background] Linnemayr S, Ryan GW, Karir V, Liu J, Palar K. Negotiation Strategies for Antiretroviral Drug Purchasers in the United States. Rand Health Q. 2012 Sep 1;2(3):7. eCollection 2012 Fall. PMID 28083266
- [Background] Linnemayr S, Ryan GW, Liu J, Palar K. Value for Money in Donor HIV Funding. Rand Health Q. 2012 Dec 1;1(4):2. eCollection 2012 Winter. PMID 28083209
- [Background] Wilson IB, Bangsberg DR, Shen J, Simoni JM, Reynolds NR, Goggin K, Gross R, Arnsten JH, Remien RH, Erlen JA, Liu H; Multisite Adherence Collaboration on HIV 14 Investigators. Heterogeneity among studies in rates of decline of antiretroviral therapy adherence over time: results from the multisite adherence collaboration on HIV 14 study. J Acquir Immune Defic Syndr. 2013 Dec 15;64(5):448-54. doi: 10.1097/QAI.0000000000000025. PMID 24225904
- [Background] Remien RH, Stirratt MJ, Dolezal C, Dognin JS, Wagner GJ, Carballo-Dieguez A, El-Bassel N, Jung TM. Couple-focused support to improve HIV medication adherence: a randomized controlled trial. AIDS. 2005 May 20;19(8):807-14. doi: 10.1097/01.aids.0000168975.44219.45. PMID 15867495
- [Background] Wagner GJ, Rabkin JG. Measuring medication adherence: are missed doses reported more accurately then perfect adherence? AIDS Care. 2000 Aug;12(4):405-8. doi: 10.1080/09540120050123800. PMID 11091773
- [Background] Arnsten JH, Demas PA, Farzadegan H, Grant RW, Gourevitch MN, Chang CJ, Buono D, Eckholdt H, Howard AA, Schoenbaum EE. Antiretroviral therapy adherence and viral suppression in HIV-infected drug users: comparison of self-report and electronic monitoring. Clin Infect Dis. 2001 Oct 15;33(8):1417-23. doi: 10.1086/323201. Epub 2001 Sep 5. PMID 11550118
- [Background] Bogart LM, Uyeda K. Community-based participatory research: partnering with communities for effective and sustainable behavioral health interventions. Health Psychol. 2009 Jul;28(4):391-3. doi: 10.1037/a0016387. PMID 19594261
- [Background] Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: assessing partnership approaches to improve public health. Annu Rev Public Health. 1998;19:173-202. doi: 10.1146/annurev.publhealth.19.1.173. PMID 9611617
- [Background] Wagner GJ, Linnemayr S, Ghosh-Dastidar B, Currier JS, Hoffman R, Schneider S. Supporting Treatment Adherence Readiness through Training (START) for patients with HIV on antiretroviral therapy: study protocol for a randomized controlled trial. Trials. 2016 Mar 24;17:162. doi: 10.1186/s13063-016-1287-3. PMID 27009061
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Smith PC, Schmidt SM, Allensworth-Davies D, Saitz R. A single-question screening test for drug use in primary care. Arch Intern Med. 2010 Jul 12;170(13):1155-60. doi: 10.1001/archinternmed.2010.140. PMID 20625025
- [Background] Bangsberg DR. Less than 95% adherence to nonnucleoside reverse-transcriptase inhibitor therapy can lead to viral suppression. Clin Infect Dis. 2006 Oct 1;43(7):939-41. doi: 10.1086/507526. Epub 2006 Aug 23. PMID 16941380
- [Background] Kobin AB, Sheth NU. Levels of adherence required for virologic suppression among newer antiretroviral medications. Ann Pharmacother. 2011 Mar;45(3):372-9. doi: 10.1345/aph.1P587. Epub 2011 Mar 8. PMID 21386024
- [Background] Shuter J, Sarlo JA, Kanmaz TJ, Rode RA, Zingman BS. HIV-infected patients receiving lopinavir/ritonavir-based antiretroviral therapy achieve high rates of virologic suppression despite adherence rates less than 95%. J Acquir Immune Defic Syndr. 2007 May 1;45(1):4-8. doi: 10.1097/QAI.0b013e318050d8c2. PMID 17460469
- [Background] Arnsten JH, Demas PA, Grant RW, Gourevitch MN, Farzadegan H, Howard AA, Schoenbaum EE. Impact of active drug use on antiretroviral therapy adherence and viral suppression in HIV-infected drug users. J Gen Intern Med. 2002 May;17(5):377-81. doi: 10.1046/j.1525-1497.2002.10644.x. PMID 12047736
- [Background] Bangsberg DR, Hecht FM, Charlebois ED, Zolopa AR, Holodniy M, Sheiner L, Bamberger JD, Chesney MA, Moss A. Adherence to protease inhibitors, HIV-1 viral load, and development of drug resistance in an indigent population. AIDS. 2000 Mar 10;14(4):357-66. doi: 10.1097/00002030-200003100-00008. PMID 10770537
- [Background] Simoni JM, Kurth AE, Pearson CR, Pantalone DW, Merrill JO, Frick PA. Self-report measures of antiretroviral therapy adherence: A review with recommendations for HIV research and clinical management. AIDS Behav. 2006 May;10(3):227-45. doi: 10.1007/s10461-006-9078-6. PMID 16783535
- [Background] Golin CE, Liu H, Hays RD, Miller LG, Beck CK, Ickovics J, Kaplan AH, Wenger NS. A prospective study of predictors of adherence to combination antiretroviral medication. J Gen Intern Med. 2002 Oct;17(10):756-65. doi: 10.1046/j.1525-1497.2002.11214.x. PMID 12390551
- [Background] Walsh JC, Mandalia S, Gazzard BG. Responses to a 1 month self-report on adherence to antiretroviral therapy are consistent with electronic data and virological treatment outcome. AIDS. 2002 Jan 25;16(2):269-77. doi: 10.1097/00002030-200201250-00017. PMID 11807312
- [Background] Buscher A, Hartman C, Kallen MA, Giordano TP. Validity of self-report measures in assessing antiretroviral adherence of newly diagnosed, HAART-naive, HIV patients. HIV Clin Trials. 2011 Sep-Oct;12(5):244-54. doi: 10.1310/hct1205-244. PMID 22180522
- [Background] Berg KM, Wilson IB, Li X, Arnsten JH. Comparison of antiretroviral adherence questions. AIDS Behav. 2012 Feb;16(2):461-8. doi: 10.1007/s10461-010-9864-z. PMID 21181252
- [Background] Sayles JN, Hays RD, Sarkisian CA, Mahajan AP, Spritzer KL, Cunningham WE. Development and psychometric assessment of a multidimensional measure of internalized HIV stigma in a sample of HIV-positive adults. AIDS Behav. 2008 Sep;12(5):748-58. doi: 10.1007/s10461-008-9375-3. Epub 2008 Apr 4. PMID 18389363
- [Background] Earnshaw VA, Quinn DM, Kalichman SC, Park CL. Development and psychometric evaluation of the Chronic Illness Anticipated Stigma Scale. J Behav Med. 2013 Jun;36(3):270-82. doi: 10.1007/s10865-012-9422-4. Epub 2012 Apr 13. PMID 22526525
- [Background] Bogart LM, Thorburn S. Are HIV/AIDS conspiracy beliefs a barrier to HIV prevention among African Americans? J Acquir Immune Defic Syndr. 2005 Feb 1;38(2):213-8. doi: 10.1097/00126334-200502010-00014. PMID 15671808
- [Background] Catz SL, Kelly JA, Bogart LM, Benotsch EG, McAuliffe TL. Patterns, correlates, and barriers to medication adherence among persons prescribed new treatments for HIV disease. Health Psychol. 2000 Mar;19(2):124-33. PMID 10762096
- [Background] Napper LE, Fisher DG, Johnson ME, Wood MM. The reliability and validity of drug users' self reports of amphetamine use among primarily heroin and cocaine users. Addict Behav. 2010 Apr;35(4):350-4. doi: 10.1016/j.addbeh.2009.12.006. Epub 2009 Dec 16. PMID 20053503
- [Background] Cherpitel CJ. Screening for alcohol problems in the U.S. general population: comparison of the CAGE, RAPS4, and RAPS4-QF by gender, ethnicity, and service utilization. Rapid Alcohol Problems Screen. Alcohol Clin Exp Res. 2002 Nov;26(11):1686-91. doi: 10.1097/01.ALC.0000036300.26619.78. PMID 12436057
- [Background] Galvan FH, Collins RL, Kanouse DE, Pantoja P, Golinelli D. Religiosity, denominational affiliation and sexual behaviors among people with HIV in the United States. J Sex Res. 2007 Feb;44(1):49-58. doi: 10.1080/00224490709336792. PMID 17599264
- [Background] Heitzmann CA, Kaplan RM. Assessment of methods for measuring social support. Health Psychol. 1988;7(1):75-109. doi: 10.1037//0278-6133.7.1.75. PMID 3277843
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Dang Q, Mazumdar S, Houck PR. Sample size and power calculations based on generalized linear mixed models with correlated binary outcomes. Comput Methods Programs Biomed. 2008 Aug;91(2):122-7. doi: 10.1016/j.cmpb.2008.03.001. Epub 2008 May 6. PMID 18462826
- [Background] Mackinnon DP, Lockwood CM, Williams J. Confidence Limits for the Indirect Effect: Distribution of the Product and Resampling Methods. Multivariate Behav Res. 2004 Jan 1;39(1):99. doi: 10.1207/s15327906mbr3901_4. PMID 20157642
- [Background] Garber AM, Phelps CE. Economic foundations of cost-effectiveness analysis. J Health Econ. 1997 Feb;16(1):1-31. doi: 10.1016/s0167-6296(96)00506-1. PMID 10167341
- [Background] Campbell MK, Torgerson DJ. Bootstrapping: estimating confidence intervals for cost-effectiveness ratios. QJM. 1999 Mar;92(3):177-82. doi: 10.1093/qjmed/92.3.177. PMID 10326078
- [Background] Gorsky RD. A method to measure the costs of counseling for HIV prevention. Public Health Rep. 1996;111 Suppl 1(Suppl 1):115-22. PMID 8862166
- [Background] Centers for Disease Control and Prevention. Complete Listing of Medication Adherence Evidence-based Behavioral Interventions. 2015; Available at: http://www.cdc.gov/hiv/research/interventionresearch/compendium/ma/complete.html.
- [Background] Results from the 2013 National Survey on Drug Use and Health: Summary of National Findings. Available at: http://www.samhsa.gov/data/sites/default/files/NSDUHresultsPDFWHTML2013/Web/NSDUHresults2013.pdf.
- [Background] Thorn B, Tadler C, Huret N, et al. WIC Participant and Program Characteristics 2014. Prepared by Insight Policy Research under Contract No. AG-3198-C-11-0010. Alexandria, VA: U.S. Department of Agriculture, Food and Nutrition Service. Available at: http://www.fns.usda.gov/sites/default/files/ops/WICPC2014.pdf;2015.
- [Background] Truman JL, Langton L. Criminal Victimization, 2014. U.S. Department of Justice, Office of Justice Programs. Available at: http://www.bjs.gov/content/pub/pdf/cv14.pdf;2015.
- [Background] LifeWindows Project Team. The LifeWindows Information Motivation Behavioral Skills ART adherence questionnaire (LW-IMB-AAQ). 2006; http://www.chip.uconn.edu/int/F_LWIMBARTQuestionnaire.pdf.
- [Background] MacKinnon DP, Lockwood CM, Williams J. Predicted and observed power rates. 2004; Available at: http://ripl.faculty.asu.edu/wp-content/uploads/2013/01/MacKinnon-Lockwood-Williams-2004-Pred-and-Obs-Power-Rates.pdf. Accessed February 7, 2014.
- [Derived] Bogart LM, Lawrence SJ, Beck A, Mutchler MG, Ball A, Thomas D, Carlisle NA, Lee DP, Nichols LL, Smith T, Wagner GJ, Goggin K, MacCarthy S. Community expert insights on anticipated implementation challenges for an evidence-based adherence intervention for Black clients. Discov Public Health. 2025;22(1):542. doi: 10.1186/s12982-025-00960-5. Epub 2025 Sep 14. PMID 40959215
- [Derived] Bogart LM, Mutchler MG, Goggin K, Ghosh-Dastidar M, Klein DJ, Saya U, Linnemayr S, Lawrence SJ, Tyagi K, Thomas D, Gizaw M, Bailey J, Wagner GJ. Randomized Controlled Trial of Rise, A Community-Based Culturally Congruent Counseling Intervention to Support Antiretroviral Therapy Adherence Among Black/African American Adults Living with HIV. AIDS Behav. 2023 May;27(5):1573-1586. doi: 10.1007/s10461-022-03921-0. Epub 2022 Nov 18. PMID 36399252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started on January 23, 2018 (and lasted until July 2020). The study setting was a large community-based HIV services organization that is connected to a Federally Qualified Health Center (FQHC) in Los Angeles County, California.
Pre-assignment Details: Prior to randomization (group assignment), 61 dropped out of the study: 51 were lost to follow-up (could not be re-contacted for randomization visit), 6 were administratively withdrawn (2 relocated out of Los Angeles, 2 died, 2 misrepresented themselves and were not Black/African American) and 4 self-withdrew (3 due to COVID-19, 1 for personal reasons).
Period: Overall Study
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
Started | 122 | 123
Completed | 85 | 81
Not Completed | 37 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rise - Treatment Education | Control - No Treatment Education | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 111 | 114 | 225
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.09 (12.38) | 48.85 (11.99) | 48.97 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 97 | 100 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 111 | 112 | 223
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 112 | 110 | 222
  White | 0 | 0 | 0
  More than one race | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 122 | 123 | 245
Continuous Adherence [Mean (Standard Deviation); unit: percentage of doses taken] — Percentage of prescribed doses that were taken during the month between baseline and the start of the intervention period Population: Adherence data, collected when participants brought in electronically monitored pill bottle caps (MEMS), was missing for some participants and some time points. Here we present all adherence data collected at baseline. Note that analysis for intervention efficacy was restricted to participants with adherence data at (a) baseline and (b) at least one of the 6 post-intervention months
  percentage of doses taken
    number analyzed (Participants) | 114 | 116 | 230
    (all) | 74.7 (22.0) | 75.7 (24.8) | 75.2 (23.4)
Dichotomous Adherence [Count of Participants; unit: Participants] — Count of participants for whom the electronically monitored percentage of prescribed dosages taken exceeded 75% during the month between baseline and the start of the intervention period Population: Adherence data, collected when participants brought in electronically monitored pill bottle caps (MEMS), was missing for some participants and some time points. Here we present all adherence data collected at baseline. Note that analysis for intervention efficacy was restricted to participants with adherence data at (a) baseline and (b) at least one of the 6 post-intervention months
  Participants
    number analyzed (Participants) | 114 | 116 | 230
    (all) | 64 | 76 | 140
Viral Suppression [Count of Participants; unit: Participants] — Viral load undetectable per venipuncture or medical records Population: Data are missing for participants who could not get venipuncture and for whom we were unable to acquire medical records (mainly b/c of COVID-19 pandemic). Here we present all data among participants with data within 6 months before baseline to 3 months after baseline (for controls) or start of intervention.
  Participants
    number analyzed (Participants) | 101 | 110 | 211
    (all) | 82 | 91 | 173
Internalized HIV Stigma [Count of Participants; unit: Participants] — Count of participants who "slightly agree" or "strongly agree" with either "Most people with AIDS are responsible for having their illness" or "A person with AIDS must have done something wrong and deserves to be punished" Population: Some responses to these questions are missing, either due to item or unit nonresponse. Here we present all collected baseline data. Note that analysis of intervention efficacy was restricted to participants with data at (a) baseline and (b) at either of the two follow-up surveys.
  Participants
    number analyzed (Participants) | 119 | 123 | 242
    (all) | 33 | 32 | 65
Medical Mistrust (HIV conspiracy beliefs) [Mean (Standard Deviation); unit: units on a scale] — Mean agreement with 9 HIV-related conspiracy beliefs. Agreement is measured on a 5-point scale from 1=Strongly Disagree to 5=Strongly Agree Population: Some responses to these questions are missing, either due to item or unit nonresponse. Here we present all collected baseline data. Note that analysis of intervention efficacy was restricted to participants with data at (a) baseline and (b) at either of the two follow-up surveys.
  units on a scale
    number analyzed (Participants) | 119 | 123 | 242
    (all) | 2.75 (0.92) | 2.59 (0.92) | 2.67 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Adherence
Description: Percentage of doses taken of those prescribed from electronic monitoring. Here we present all data collected at all time points used in analysis. Evaluation of intervention efficacy was performed with repeated measures regression using continuous adherence measurements at all 6 months post-intervention (7th through 12th month post-baseline) and was restricted to those with adherence data at baseline.
Time Frame: baseline (pre-treatment) and post-treatment observations at 7, 8, 9, 10, 11, and 12 months post-baseline
Population: Adherence data, collected when participants brought in electronically monitored pill bottle caps (MEMS), was missing for some participants and some time points. As can be seen below, the # of participants with adherence data varies by time point; the numbers above are the total number of participants included in the analysis (adherence data present at baseline and at least one follow-up time point)
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
Number analyzed (Participants) | 83 | 81
percentage of doses taken
  7 months post-baseline: number analyzed (Participants) | 80 | 78
  7 months post-baseline | 68.80 (29.63) | 70.95 (27.24)
  8 months post-baseline: number analyzed (Participants) | 73 | 76
  8 months post-baseline | 72.76 (26.16) | 70.02 (26.11)
  9 months post-baseline: number analyzed (Participants) | 71 | 76
  9 months post-baseline | 72.09 (25.39) | 64.62 (31.41)
  10 months post-baseline: number analyzed (Participants) | 72 | 63
  10 months post-baseline | 71.27 (27.59) | 71.08 (25.24)
  11 months post-baseline: number analyzed (Participants) | 71 | 67
  11 months post-baseline | 69.87 (28.26) | 63.76 (31.44)
  12 months post-baseline: number analyzed (Participants) | 63 | 58
  12 months post-baseline | 70.32 (26.77) | 70.46 (23.55)
Statistical Analysis 1: Comparison: Rise - Treatment Education vs Control - No Treatment Education; Tested with repeated measures linear regression where all 6 past-month post-intervention measurements of adherence were stacked together such that each participant could contribute up to 6 records. Standard errors were adjusted for clustering on participant, and weights for presence of data were used. Fixed effects were an intervention indicator and continuous adherence measured at baseline. Model included all participants with adherence data (a) at baseline and (b) at least one follow-up month; Test type: Superiority; p = .08, Regression, Linear; Model is adjusted for participant sex, which was found to be significantly associated with adherence in a similar repeated measures model; Mean Difference (Net) = 6.89, 95% CI 2-sided [-0.82 to 14.61], Standard Error of Mean 3.91 — Values entered are for regression coefficient for intervention indicator (versus control) and represents the adjusted difference across all follow-up time points

2. Primary Outcome: Dichotomous Adherence
Description: Number of Participants who Reported Taking Greater Than or Equal to 75% of Prescribed Dosage, based on electronic monitoring. Here we present all data collected at all time points used in analysis. Evaluation of intervention efficacy was performed with repeated measures regression using adherence measurements at all 6 months post-intervention (7th through 12th month post-baseline) and was restricted to those with adherence data at baseline.
Time Frame: baseline (pre-treatment) and post-treatment observations at 7, 8, 9, 10, 11, and 12 months post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
Number analyzed (Participants) | 83 | 81
Participants
  7 months post-baseline: number analyzed (Participants) | 80 | 78
  7 months post-baseline | 45 | 43
  8 months post-baseline: number analyzed (Participants) | 73 | 76
  8 months post-baseline | 44 | 40
  9 months post-baseline: number analyzed (Participants) | 71 | 76
  9 months post-baseline | 43 | 38
  10 months post-baseline: number analyzed (Participants) | 72 | 63
  10 months post-baseline | 42 | 32
  11 months post-baseline: number analyzed (Participants) | 71 | 67
  11 months post-baseline | 40 | 29
  12 months post-baseline: number analyzed (Participants) | 63 | 58
  12 months post-baseline | 37 | 28
Statistical Analysis 1: Comparison: Rise - Treatment Education vs Control - No Treatment Education; Tested with repeated measures logistic regression where all 6 past-month post-intervention measurements of adherence were stacked together such that each participant could contribute up to 6 records. Standard errors were adjusted for clustering on participant, and weights for presence of data were used. Fixed effects were an intervention indicator and baseline dichotomous adherence. Model included all participants with adherence data (a) at baseline and (b) at least one follow-up month; Test type: Superiority; p = .0257, Regression, Logistic — Per above, p-value is from repeated measures logistic regression with standard errors adjusted for clustering on participant; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.09 to 3.60] — Odds ratio is for intervention indicator (versus controls)

3. Primary Outcome: Viral Suppression
Description: Viral load undetectable per venipuncture or medical records
Time Frame: baseline (pre-treatment) and post-treatment observations at 7 and 12 months post-baseline. For 7M, medical records were used if within 90 days of survey completion; for 13 months, medical records were used if within 90 days before or 180 days after survey
Population: Data are missing for participants who were unable to come in for venipuncture and for whom we were unable to acquire medical records within 90 days of the 7-month survey OR within 90 days before / 180 days after 13 month survey. As can be seen below, the # of participants with adherence data varies by time point; the numbers above are the total number of participants included in the analysis (data present at baseline and at either follow-up time point).
Measure: Count of Participants; unit: Participants
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
Number analyzed (Participants) | 68 | 83
Participants
  7 month post-baseline: number analyzed (Participants) | 51 | 72
  7 month post-baseline | 45 | 60
  12 month post-baseline: number analyzed (Participants) | 55 | 63
  12 month post-baseline | 50 | 56
Statistical Analysis 1: Comparison: Rise - Treatment Education vs Control - No Treatment Education; Tested with repeated measures logistic regression where both post-intervention measurements were stacked together such that each participant could contribute up to 2 records. Standard errors were adjusted for clustering on participant, and weights for presence of viral suppression data were used. Fixed effects were an intervention indicator and baseline viral suppression. Model included all viral suppression data (a) at baseline and (b) close to either of the two follow-up surveys; Test type: Superiority; p = .26, Regression, Logistic — As mentioned above, p-value comes from repeated measures regression with standard errors adjusted for clustering on participant; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.64 to 5.18] — Odds ratio is for intervention indicator (versus controls)

4. Secondary Outcome: Internalized HIV Stigma
Description: Measure is count of participants who "slightly agree" or "strongly agree" with either "Most people with AIDS are responsible for having their illness" or "A person with AIDS must have done something wrong and deserves to be punished."
Time Frame: baseline (pre-treatment) and post-treatment observations at 7 and 12 months post-baseline
Population: Data may be missing due to unit or item nonresponse. As can be seen below, the # of participants with stigma data varies by time point; the numbers above are the total number of participants included in the analysis (data present at baseline and at either follow-up time point)
Measure: Count of Participants; unit: Participants
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
Number analyzed (Participants) | 94 | 96
Participants
  7 months post-baseline: number analyzed (Participants) | 85 | 87
  7 months post-baseline | 25 | 29
  12 months post-baseline: number analyzed (Participants) | 83 | 80
  12 months post-baseline | 15 | 26
Statistical Analysis 1: Comparison: Rise - Treatment Education vs Control - No Treatment Education; Tested with repeated measures logistic regression where both post-intervention responses were stacked together such that each participant could contribute up to 2 records. Standard errors were adjusted for clustering on participant, and weights for follow-up response were used. Fixed effects were an intervention indicator and baseline stigma. Model included all participants with responses (a) at baseline and (b) at least one of the two follow-up surveys; Test type: Superiority; p = .05, Regression, Logistic — As mentioned above, p-value is from repeated measures regression with standard errors adjusted for clustering on participant; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.32 to 1.00] — Odds ratio is for intervention indicator (versus controls)

5. Secondary Outcome: Medical Mistrust
Description: Outcome is mean agreement with 9 HIV-related conspiracy beliefs, each measured on a 5-point scale from 1=Strongly Disagree to 5=Strongly Agree.
Time Frame: baseline (pre-treatment) and post-treatment observations at 7 and 12 months post-baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
Number analyzed (Participants) | 94 | 97
score on a scale
  7 months post-baseline: number analyzed (Participants) | 85 | 88
  7 months post-baseline | 2.62 (1.04) | 2.65 (0.92)
  12 months post-baseline: number analyzed (Participants) | 83 | 81
  12 months post-baseline | 2.41 (0.94) | 2.56 (1.07)
Statistical Analysis 1: Comparison: Rise - Treatment Education vs Control - No Treatment Education; Tested with repeated measures linear regression where both post-intervention responses were stacked together such that each participant could contribute up to 2 records. Standard errors were adjusted for clustering on participant, and weights for follow-up response were used. Fixed effects were an intervention indicator and baseline stigma. Model included all participants with responses (a) at baseline and (b) at least one of the two follow-up surveys; Test type: Superiority; p = .0199, Regression, Linear — As described above, p-value is from repeated measures regression with standard errors adjusted for clustering on participant; Mean Difference (Net) = -0.215, 95% CI 2-sided [-0.395 to -0.034], Standard Error of Mean 0.091 — Estimation parameter is the regression coefficient for intervention indicator (vs. control) and represents the adjusted difference across both follow-up time points

ADVERSE EVENTS:
Time Frame: 12 months (the timeframe that each participant was in the study)
Description: The definition did not differ
Arm/Group | Rise - Treatment Education | Control - No Treatment Education
All-Cause Mortality (participants affected / at risk) | 0/122 | 2/123
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/123
Other Adverse Events (participants affected / at risk) | 3/122 | 3/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rise - Treatment Education (N=122) | Control - No Treatment Education (N=123)
Other Adverse Event (General disorders) | 3 (3) | 3 (3) — Includes hospitalizations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03331978/Prot_003.pdf
  • Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03331978/SAP_004.pdf
  • Informed Consent Form (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03331978/ICF_005.pdf